CLINICAL TRIAL: NCT04933383
Title: A Prospective, Active-controlled, Randomized, Open Label, Single-center, Multiple Dose, Crossover Clinical Trial to Assess the Efficacy, Safety and PK of AQ001S Compared to a Budesonide Inhalation Suspension in Adults With Mild Asthma
Brief Title: Crossover Trial to Assess Efficacy and Safety of Inhaled AQ001S Compared to a Budesonide Suspension in Mild Asthmatics
Acronym: BOREAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aquilon Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AQ-PRO-005
Record Dates: First submitted 2021-05-31; First posted 2021-06-21 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AQ001S 0.125 mg/ml (Experimental): AQ001S 0.125 mg/ml is a budesonide inhalation solution administered by nebulization once daily.
  Interventions: Drug: AQ001S 0.125 mg/ml; Drug: Budesonide 0.125 mg/ml inhalation suspension
- budesonide inhalation suspension 0.125 mg/ml (Active Comparator): Budesonide 0.125 mg/ml is a budesonide inhalation suspension administered by nebulization once daily.
  Interventions: Drug: AQ001S 0.125 mg/ml; Drug: Budesonide 0.125 mg/ml inhalation suspension

INTERVENTIONS:
Drug: AQ001S 0.125 mg/ml — administered by nebulization once daily
  Other Names: budesonide inhalation solution 0.125 mg/ml
Drug: Budesonide 0.125 mg/ml inhalation suspension — administered by nebulization once daily
  Other Names: Budesonide inhalation suspension 0.125 mg/ml

SUMMARY:
This is a prospective, active-controlled, randomized, open label, single-center, multiple dose, two-period crossover clinical trial to assess the efficacy, safety and pharmacokinetics of AQ001S compared to a budesonide inhalation suspension (comparator) in adults with mild asthma.

Both treatments will be administered by nebulization.

DETAILED DESCRIPTION:
Adults patients with mild asthma (18 to 65 years old), who are 'inhaled corticosteroid (ICS)'-naïve for minimum 60 days at Screening Visit will be enrolled in the study. The patients will be treated for 28 days. The primary endpoint will be assessed by a provocative concentration of methacholine that results in a 20% drop (PC20) in the first second forced expiratory volume (FEV1) as determined by methacholine challenge test. The pharmacokinetics (PK) endpoint, i.e. PK profile of budesonide in plasma, and pharmacodynamics (PD) endpoints, i.e. recording of symptom scores, use of reliever drugs as needed, biomarkers of airway inflammation and pulmonary function tests will be assessed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.5 and 29 kg/m2.
* Documented clinical diagnosis of stable, persistent, asthma for at least 3 months
* Subjects who are ICS-naïve for minimum 60 days at Screening Visit.
* Positive methacholine (MCh) challenge test (concentration of MCh provoking an FEV1 fall of 20% [PC20] < 8 mg/ml or dose of MCh provoking an FEV1 fall of 20% [PD20] < 0.2 mg) in the last year.
* Post-bronchodilator FEV1 at least 80% of the predicted, documented in the last year.
* Clinical laboratory test results, 12-lead electrocardiogram (ECG), blood pressure and heart rate (supine) within normal reference range or judged to be not clinically significant by the Investigator.
* Female subjects of childbearing potential should have a negative pregnancy test at Screening Visit and use a highly effective method of contraception.
* Reliable subjects who are willing to be available for the duration of the clinical trial and willing to comply with clinical trial procedures.
* Subjects who have the ability to understand the requirements of the clinical trial.
* Subjects who have given written informed consent.

Exclusion Criteria:

* Current smokers or recent (< 8 weeks) ex-smokers or ex-smokers if > 10 pack-years.
* Pregnant or breastfeeding female subjects.
* Inability to carry out pulmonary function testing.
* FEV1 < 70%.
* History of near-fatal asthma and/or intensive care unit admission for asthma symptoms.
* Exacerbations of asthma requiring oral steroids, hospitalization or change in asthma treatment in the previous three months.
* Evidence of symptomatic chronic or acute respiratory infection in the previous 8 weeks.
* Diagnosis of chronic obstructive pulmonary disease (COPD) or bronchiectasis.
* Pulmonary malformations, tuberculosis, cystic fibrosis.
* History of hypersensitivity or existing contraindication to budesonide or any other Investigational Medicinal Product (IMP) ingredients.
* Untreated oral candidiasis.
* Immunosuppressive treatment, including systemic corticosteroids (e.g., oral, parenteral, ocular, nasal), within 28 days before Screening Visit.
* Use of ICS within 60 days before Screening Visit.
* Use of anti-leukotrienes, immunoglobulins, beta-blockers, digitalis, amiodarone, antifungals, macrolides, antidepressants, monoamine oxidase inhibitors, antiretroviral drugs, cholinesterase inhibitors, histamine, theophylline, non-steroidal anti-inflammatory drugs, anticholinergic drugs, neuroleptics, curariform drugs, antihistaminic (anti-H1) drugs, calcium channel blockers, long acting beta2-antagonists, mast cell stabilizers (e.g. natrium cromoglycate).
* History of alcohol or drug abuse.
* Unstable or life-threatening cardiac disease
* History or presence of prolonged QT interval (> 470 ms), or any other clinically significant ECG abnormalities as judged by the Investigator based on 12-lead ECG recordings at Screening Visit.
* Diabetes mellitus.
* Neuropsychiatric diseases.
* Clinically relevant laboratory abnormalities at Screening Visit.
* Blood or plasma donation within 30 days prior to Screening Visit.
* History or presence of malignancy of any system organ class (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years prior to Screening Visit, regardless of whether there is evidence of local recurrence or metastases.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the clinical trial.
* History or presence of any other clinically relevant disease of any major system organ class (e.g. cardiovascular, pulmonary, renal, hepatic, gastrointestinal, reproductive, endocrinological, neurological, psychiatric or orthopedic disease) as judged by the Investigator.
* Human immunodeficiency virus (HIV) and severe acute respiratory syndrome (SARS)-CoV-2 infections.
* Subjects who participated in an investigational trial within the 12 weeks prior to the start of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Benoît Martinot, Principal Investigator — Pneumocare SPRL
Locations (1):
- Pneumocare SPRL, Erpent, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cross-over part of the study (treatment period 1) - Washout period of 2 weeks - Cross-over part of the study (treatment period 2)
Groups:
- Sequence A: AQ001S - Comparator: AQ001S budesonide solution was administered for 29 (+2) days once daily (treatment period 1).
  Following a wash-out period of 14 (+2) days, the comparator Budesonide suspension was administered for 29 (+2) days once daily (treatment period 2).
- Sequence B: Comparator - AQ001S: The comparator Budesonide suspension was administered for 29 (+2) days once daily (treatment period 1). Following a wash-out period of 14 (+2) days, AQ001S budesonide solution was administered for 29 (+2) days once daily (treatment period 2).
Period: Overall Study
Arm/Group | Sequence A: AQ001S - Comparator | Sequence B: Comparator - AQ001S
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The efficacy population encompasses all subjects that completed both treatment periods and for which the primary efficacy parameters PC20 is available at baseline (visit 1) and after both treatment periods (visit 2 and visit 4).
  The safety population includes all randomized subjects who received at least one dose of the study medication (AQ001S or comparator).
Groups:
- Sequence A: AQ001S - Comparator: AQ001S budesonide solution was administered for 29 (+2) days once daily (treatment period 1). Following a wash-out period of 14 (+2) days, the comparator (budesonide suspension) was administered for 29 (+2) days once daily (treatment period 2).
- Sequence B: Comparator - AQ001S: The comparator (budesonide suspension) was administered for 29 (+2) days once daily (treatment period 1). Following a washout period of 14 (+2) days, AQ001S budesonide solution was administered for 29 (+2) days once daily (treatment period 2).
- Total: Total of all reporting groups
Arm/Group | Sequence A: AQ001S - Comparator | Sequence B: Comparator - AQ001S | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (11.2) | 29.1 (9.9) | 32.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 11 | 12 | 23
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 24.38 (2.91) | 24.24 (3.86) | 24.31 (3.36)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PC20 After Each Treatment Period Assessed by Methacholine (MCh) Challenge Test
Description: At Visit 1 (baseline), Visit 2 (29-day treatment period 1) and Visit 4 (29-day treatment period 2), a MCh challenge test will be performed, i.e. up to the administration of a concentration of MCh provoking an FEV1 fall of 20% (PC20). FEV1 is measured by spirometry. The change in PC20 from baseline to the end of each period (two periods) was assessed.
Time Frame: visit 1 (baseline) - visit 2 (at the end of Treatment Period 1) and visit 4 (end of Treatment Period 2)
Population: The efficacy population encompasses all subjects that completed both treatment periods and for which the primary efficacy parameter PC20 was available at baseline (visit 1) and after both treatment periods (visit 2 and visit 4).
Measure: Mean (95% Confidence Interval); unit: mg/mL
Groups:
- AQ001S 0.125 mg/ml: AQ001S is a budesonide inhalation solution administered by nebulization once daily.
  AQ001S 0.125 mg/ml: administered by nebulization once daily
- Budesonide Inhalation Suspension 0.125 mg/ml: The comparator is a budesonide inhalation suspension administered by nebulization once daily.
  Budesonide 0.125 mg/ml inhalation suspension: administered by nebulization once daily
Arm/Group | AQ001S 0.125 mg/ml | Budesonide Inhalation Suspension 0.125 mg/ml
Number analyzed (Participants) | 22 | 22
mg/mL | 3.7 [0.9 to 6.5] | 1.2 [-0.7 to 3.0]
Statistical Analysis 1: Comparison: AQ001S 0.125 mg/ml vs Budesonide Inhalation Suspension 0.125 mg/ml; The primary efficacy endpoint is the change from baseline in PC20 after each treatment period (baseline is defined at Visit 1). For primary efficacy analysis, the mean PC20 changes from baseline between AQ001S and the comparator were compared by analysis of covariance (ANCOVA) for crossover design. A p-value was calculated for the difference of the parameter between AQ001S and the comparator. Additionally, an adjusted 95%-CI for the mean difference was obtained by the ANCOVA; Test type: Superiority; p = 0.000813, ANCOVA; difference/ratio of least square means = 180.6, 95% CI 2-sided [106.42 to 306.48]

2. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Incidence of Treatment-Emergent Adverse Events as assessed by collection of (Serious) Adverse Events
Time Frame: Over the treatment period, from the informed consent signature up to the end of second 29-day treatment period
Population: The safety population includes all randomized subjects who received at least one dose of the study medication (AQ001S or comparator).
Measure: Number; unit: events
Groups:
- Budesonide Inhalation Suspension 0.125 mg/ml: The comparator Budesonide suspension is a budesonide inhalation suspension administered by nebulization once daily.
  Budesonide 0.125 mg/ml inhalation suspension: administered by nebulization once daily
Arm/Group | AQ001S 0.125 mg/ml | Budesonide Inhalation Suspension 0.125 mg/ml
Number analyzed (Participants) | 23 | 23
events
  All-Cause Mortality | 0 | 0
  Serious Adverse Events | 0 | 0
  Other (not including serious) Adverse Events | 3 | 10

ADVERSE EVENTS:
Time Frame: Adverse events/serious adverse events were recorded from the time the subjects signed the informed consent until the last study visit.
Arm/Group | AQ001S 0.125 mg/ml | Budesonide Inhalation Suspension 0.125 mg/ml
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 4/23 | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AQ001S 0.125 mg/ml (N=23) | Budesonide Inhalation Suspension 0.125 mg/ml (N=23)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
No limitations or caveat are reported for this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication and disclosure of results of this trial must be consistent with Aquilon Pharmaceuticals publication policy. The rights of the investigator and the sponsor with regard to publication or disclosure of the results of this trial are described in the investigator contract.

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04933383/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT04933383/SAP_001.pdf